CLINICAL TRIAL: NCT05005546
Title: The Effect of Yoga and Laughter Yoga on Increasing the Psychological Resilience of Mothers With Their Babies in the Neonatal Intensive Care Unit
Brief Title: The Effect of Yoga and Laughter Yoga on Increasing the Psychological Resilience of Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/085
Record Dates: First submitted 2021-08-07; First posted 2021-08-13 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Depression; Stress; Anxiety; Psychological Resilience
Keywords: Psychological Resilience; Depression; Stress; Anxiety; Nursing
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Yoga; Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Yoga (Experimental)
  Interventions: Behavioral: Yoga
- Experimental: Laughter Yoga (Experimental)
  Interventions: Behavioral: Laughter Yoga
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Yoga — Yoga will be applied to mothers in the yoga group
  Arms: Experimental: Yoga
Behavioral: Laughter Yoga — Laughter Yoga will be applied to mothers in the yoga group
  Arms: Experimental: Laughter Yoga

SUMMARY:
Objective: The study will carried out in a randomized controlled trial to determine the effect of yoga and laughter yoga on increasing the psychological resilience of mothers with their babies in the Neonatal Intensive Care Unit

Method: The research will be carried out with mothers whose babies are treated in the neonatal intensive care unit. Mothers will be divided into three groups as yoga (n=20), laughter yoga (n=20) and control (n=20) by block randomization method. Research findings; Data Form will obtained by using "Introductory Characteristics Form", "Depression, Anxiety, Stress Scale (DASS-21)" and "Psychological Resilience Scale".

DETAILED DESCRIPTION:
Starting from the 1st week (5-7 days) after the birth, mothers will be given 10 sessions of laughter yoga (laughter group) and yoga (yoga group) twice a week for 45 minutes.DASS-21 and Resilience Scale will be administered to mothers in all groups at 1st, 3rd and 5th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are older than 18 years of age,
* whose gestational week is less than 32 weeks,
* whose baby has been treated in the neonatal intensive care unit for at least one week,
* who have internet access

Exclusion Criteria:

* Mothers with a genetic disease or congenital anomaly in their baby

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety, Stress Scale (DASS-21) | 0-3 point each item, min 0-max 21 total point each subscale
  It is an assessment tool developed to evaluate the depression, anxiety and stress levels of individuals.
Psychological Resilience Scale | min 0-max 40 point
  The scale is a scale developed to determine the psychological resilience of individuals, which enables them to return to their former state after negative events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol